CLINICAL TRIAL: NCT00460356
Title: Glycoprotein and Glycan Profiling in Patients With Locally Advanced Cervical Cancer (Stage IB2, IIA > 4 CM, IIB to IVA) Undergoing Pelvic and Para-aortic (Abdominal) Lymphadenectomy
Brief Title: Glycoprotein and Glycan in Tissue and Blood Samples of Patients With Stage IB-IVA Cervical Cancer Undergoing Surgery to Remove Pelvic and Abdominal Lymph Nodes
Status: Completed | Type: Observational
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: GOG Foundation (Network)
Other Study IDs: GOG-0221; NCI-2009-00592 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000540243; GOG-0221 (Other: NRG Oncology); GOG-0221 (Other: CTEP); U10CA180868 (NIH); U10CA027469 (NIH)
Record Dates: First submitted 2007-04-11; First posted 2007-04-13 (Estimated); Last update posted 2017-08-24 (Actual); Status verified 2017-08

CONDITIONS: Cervical Adenocarcinoma; Cervical Adenosquamous Carcinoma; Cervical Small Cell Carcinoma; Cervical Squamous Cell Carcinoma, Not Otherwise Specified; Stage IB Cervical Cancer; Stage IIA Cervical Cancer; Stage IIB Cervical Cancer; Stage III Cervical Cancer; Stage IVA Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Lymph Node Excision

GROUPS / COHORTS (1):
- Ancillary-Correlative (glycoprotein and glycan profiling): Primary and metastatic tumor specimens are collected during lymphadenectomy and used for tissue microarray analysis, mutational analysis of T-synthase and Cosmc, immunohistochemical staining of Tn antigen and sialyl Tn antigen, and customized gene expression array analysis of 400 genes associated with glycobiology. Pre-lymphadenectomy blood is collected from patients at baseline for customized glycan array analysis of 300 carbohydrates.
  Interventions: Other: Laboratory Biomarker Analysis; Procedure: Lymphadenectomy

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Procedure: Lymphadenectomy — Undergo lymphadenectomy
  Other Names: excision of the lymph node; lymph node dissection; lymph node excision

SUMMARY:
This clinical trial studies glycoprotein and glycan in tissue and blood samples of patients with stage IB-IVA cervical cancer undergoing surgery to remove pelvic and abdominal lymph nodes. Studying samples of tumor tissue and blood from patients with cancer in the laboratory may help doctors learn more about changes that occur in deoxyribonucleic acid (DNA) and identify biomarkers related to cancer. It may also help doctors learn how far the disease has spread.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Determine whether the presence of a mutation in T-synthase or Cosmc and/or the presence of positive immunohistochemical expression of Tn antigen or sialyl Tn antigen in tumor specimens is associated with progression-free or overall survival in patients with stage IB2, II, III, or IVA cervical cancer undergoing pelvic and para-aortic (abdominal) lymphadenectomy.

SECONDARY OBJECTIVES:

I. Determine whether the presence of a mutation in T-synthase or Cosmc and/or the presence of positive immunohistochemical expression of Tn antigen or sialyl Tn antigen in tumor specimens is associated with lymph node metastasis or local control.

II. Identify a glycoprotein profile from a customized gene expression array analysis in tumor specimens or a glycan profile from a customized glycan array in serum that is associated with lymph node metastasis, local control, disease recurrence/progression, or survival.

III. Determine whether differences exist in T-synthase or Cosmc mutations, the immunohistochemical expression of Tn antigen or sialyl Tn antigen, and glycoprotein profiling (using customized gene expression array analysis) in matched primary tumor compared with metastatic lymph nodes that are associated with lymph node metastasis, local control, disease recurrence/progression, or survival.

IV. Identify differences in glycoprotein expression profiling and glycan profiling in tumor specimens with or without a mutation in T-synthase or Cosmc, or in tumor specimens with or without positive immunohistochemical expression of Tn antigen or sialyl Tn antigen that are associated with lymph node metastasis, local control, disease recurrence/progression, or survival.

OUTLINE:

Primary and metastatic tumor specimens are collected during lymphadenectomy and used for tissue microarray analysis, mutational analysis of T-synthase and Cosmc, immunohistochemical staining of Tn antigen and sialyl Tn antigen, and customized gene expression array analysis of 400 genes associated with glycobiology. Pre-lymphadenectomy blood is collected from patients at baseline for customized glycan array analysis of 300 carbohydrates.

After completion of study treatment, patients are followed up every 3 months for 2 years and then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients with primary, previously untreated, histologically confirmed locoregionally advanced (Stages IB2, IIA > 4 cm, IIB-IVA) invasive carcinoma of the cervix (any cell type) who will undergo pelvic and para-aortic (abdominal) lymphadenectomy to determine the presence or absence of lymph node metastasis
* Patients who have met the pre-entry requirements
* Patients with a block or 25 unstained sections of formalin-fixed and paraffin-embedded primary tumor available to satisfy the primary tumor requirement
* Patients who have signed an approved informed consent and authorization permitting release of personal health information

Exclusion Criteria:

* Patients who do not satisfy pre-entry requirements

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Sampling Method: Probability Sample
Enrollment: 159 (Actual)
Dates: Start 2007-04-02 (Actual); Primary Completion 2016-07-16 (Actual); Study Completion 2016-07-16 (Actual)

PRIMARY OUTCOMES:
Differences in 10 of the 300 carbohydrates under examination using the customized glycan array | Up to 3 years
Differences in approximately 50 of the 400 genes on the customized glycogene expression array | Up to 3 years
Level of immunohistochemical staining for Tn antigen and sialyl Tn antigen | Up to 3 years
Presence of T-synthase or Cosmc mutation | Up to 3 years

SECONDARY OUTCOMES:
Local control | Up to 3 years
Lymph node metastasis | Up to 3 years
Overall survival | Up to 3 years
Progression-free survival (recurrence and disease progression) | Up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Michael Gold, Principal Investigator — NRG Oncology
Locations (18):
- United States (18):
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Olive View-University of California Los Angeles Medical Center, Sylmar, California
  - Augusta University Medical Center, Augusta, Georgia
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Saint Louis University Hospital, St Louis, Missouri
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - Women's Cancer Center of Nevada, Las Vegas, Nevada
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Summa Akron City Hospital/Cooper Cancer Center, Akron, Ohio
  - University of Cincinnati/Barrett Cancer Center, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - Lake University Ireland Cancer Center, Mentor, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Women and Infants Hospital, Providence, Rhode Island